CLINICAL TRIAL: NCT04735601
Title: Ahmed Valve Implantation Coated With Poly Lactic -Co-glycolic Acid (PLGA) Saturated With Mitomycin-C in the Management of Adult Onset Glaucoma in Sturge Weber Syndrome
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Hany Mahmoud, principal investigator, Sohag University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S20-161
Record Dates: First submitted 2021-01-23; First posted 2021-02-03 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ahmed valve coated with PLGA is implanted in secondary glaucoma in Sturge Weber syndrome (Experimental): Ahmed valve coated with PLGA is implanted in secondary glaucoma in Sturge Weber syndrome
  Interventions: Procedure: Ahmed Valve
- Ahmed valve implanted in secondary glaucoma in Sturge Weber syndrome (Active Comparator): Ahmed valve will be implanted alone with no PLGA
  Interventions: Procedure: Ahmed Valve

INTERVENTIONS:
Procedure: Ahmed Valve — Ahmed valve implantation coated with poly lactic -co-glycolic acid (PLGA) saturated with Mitomycin-C in the management of adult onset glaucoma in Sturge Weber syndrome

SUMMARY:
Sturge weber's syndrome is an oculcutaneous syndrome, ocular manifestations may include heamangioma in the eye lids, choroidal heamangioma, or glaucoma, the glaucoma may present at infancy and may be due to resistance to aqueous outflow through trabecular meshwork(1), it may develop later and this is due to episcleral venous raised pressure.(2-3) Glaucoma associated with Sturge weber syndrome is difficult to be treated medically with high risk of complications when treated with bleb -based surgeries. Suprachoroidal hemorrhage or detachment is a challenging complication which must be encountered.

The usage of Ahmed valve in the management of glaucoma associated with Sturge weber syndrome is a bleb based procedure carries the risks of over filtration or encapsulation and decreased filtration with failure to control glaucoma.

The use of Ahmed valve in the management of pediatric glaucoma associated with Sturge weber syndrome has better results as recorded by Nassiri et al. Ahmed valve implantation can have some drawbacks such as pupillary irregularity, lens opacification, or encapsulation.(4-7) Glaucoma drainage devices such as Ahmed valve, Molteno or Braeveldt valve can be used when other methods of treatment fail, they provide alternative pathway to the aqueous to be collected in a plate positioned under the conjunctiva, (8-10) Encapsulation is a major problem occurs around the end plate due to fibrous reaction and so the drainage of the aqueous is decreased , Epatein (11) attributed that to fibro vascular proliferation in the episcleral tissue .the fibrous reaction is multifactorial , it may be due to the size of the end plate, the biomaterial, design or the shape of the plate.

The use of drainage devices with advanced drug delivery system can improve the success of drainage device.

A double-layered porous coating for Ahmed glaucoma valves based on biodegradable poly(lactic-co-glycolic acid) (PLGA) was described by Ponnusamy et al. [12] to produce continuous release of antifibrotic agents [mitomycin C (MMC) and/or 5-fluorouracil (5-FU)] to the subconjunctival space. This release continue for about one month with decreasing fibrosis, the nanofiltration membrane could entrap the proteins passing out from the anterior chamber leading to minimal increase in aqueous resistance.(12-13)

DETAILED DESCRIPTION:
All participants will be evaluated regarding the following:

Visual acuity (VA) will be measured before and after surgery. Visual field (VF) will be assessed. Optical coherence topography (OCT) Ahmed valve coated with PLGA nanoparticles saturated with Mitomycin-C 2mg/ml. Follow up will continue for one year regarding intraocular pressure IOP, VA , VF, OCT and occurrence of complications such as erosion, extrusion, infection, encapsulation and fibrosis around the stent.

Data will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffered from adult onset Sturge Weber syndrome and subjected to Ahmed valve implantation.

Exclusion Criteria:

* other ocular pathology; choroidal heamangioma, cataract, exudative retinal detachment.

Patients under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2022-12-15 (Estimated)

PRIMARY OUTCOMES:
IOP in mmg | one year
  efficacy of Ahmed valve implantation coated with PLGA sturated with MMC
Incidence of complications | one year
  to assess complications regarding the flap , erosions to the conjunctiva , extrusion , endothelial toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Hany Mahmoud, MD, Principal Investigator — Sohag University
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: one year